CLINICAL TRIAL: NCT04407897
Title: SOFT - A Phase 2 Study of Stereotactic Ablative Radiotherapy of Infra-diaphragmatic Soft Tissue Metastases
Brief Title: SOFT- Stereotactic Ablative Radiotherapy of Infra-diaphragmatic Soft Tissue Metastases
Acronym: SOFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Henry Ford Hospital (Other)
Responsible Party: Principal Investigator, Mette Felter, Principal Investigator, MD, Mette Felter, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-19014486
Record Dates: First submitted 2020-05-17; First posted 2020-05-29 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor; Oligometastases; Soft Tissue Disease
Keywords: SBRT; SABR; MR-guided radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is a prospective investigator-initiated phase II multicentre-study, investigating the toxicity and efficacy of SABR for infra-diaphragmatic tumors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Experimental): Patients with oligometastatic lesions, fulfilling the inclusion/exclusion criteria's will be assigned to SABR.
  Interventions: Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Three different dose fractionation schemes will be available: 45 Gy in 3 fractions, 50 Gy in 5 fractions, and 60 Gy in 8 fractions.

SUMMARY:
The SOFT study will evaluate the feasibility and safety of MR-guided stereotactic ablative radiotherapy (SABR) for infra-diaphragmatic soft tissue metastases.

DETAILED DESCRIPTION:
The investigators wish to evaluate the safety and feasibility of MR-guided stereotactic radiation to patients with infra-diaphragmatic oligometastatic disease including quality of life assessments and patient-reported outcome measures. Further, the investigators assess clinical response among patients with oligometastatic disease (OMD), defined as up to five metastases in up to three different organs.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytology proven non-haematological cancer.
* At least one metastasis should be localized in the infra-diaphragmatic soft tissue.
* Eastern Cooperative Oncology Group (ECOG) scale of performance status ≤ 2.
* ≥ 18 years old.
* Life expectancy > 6 months.
* Target diameter (GTV) ≤ 5 cm.
* Metastatic lesions must be visible, imaging defined targets and suitable for treatment with SABR.
* In case of de novo OMD and oligometastatic recurrence a maximum of 5 targets (including the primary tumour) in a maximum of 3 organ sites are allowed.
* In case of oligoprogressive disease (OPD) * and induced OMD ** only 3 metastases (including the primary tumour) are allowed.
* All metastatic sites are treated or planned for ablative therapy (including surgery). For OPD, only the sites in progression is required to fulfil this criterion.
* A baseline scan within 28 days of inclusion (PET-CT or CT and MR scanning).
* No curative intended treatment option available.
* An ablative strategy should be deemed clinically relevant and it is at the discretion of the treating physician to decide.
* Ability to understand and the willingness to sign a written informed consent document.
* If the target is in the liver, a Child-Pugh Score A is required.

Exclusion Criteria:

* Patient cannot tolerate physical set up required for SABR.
* Active bowel obstruction.
* Uncontrolled intercurrent illness.
* Medical contraindication to undergoing MR-imaging.
* Pregnancy.
* Patients with uncontrolled brain metastases.
* Uncontrolled disease in respect to malignant pleural effusion, ascites, lymphangitic carcinomatosis, pleural carcinomatosis or peritoneal carcinomatosis.
* If the patient has received previous radiotherapy, the combined dose at the radiation site must not exceed the dose constraints.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative CTCAE grade ≥ 4 SABR related toxicity (TRAE). | Assessed at 1 year.
  Registration of toxicity will be assessed according to a prespecified selection of organ related adverse events defined by CTCAE version 5.0.

SECONDARY OUTCOMES:
Freedom from local progression. | Assessed at week 6, 12, 24, 36, and 52.
  Defined as the time from inclusion to local progression as determined by investigator using RECIST 1.1 criteria.
Progression free survival. | Assessed at week 6, 12, 24, 36, and 52.
  The time from inclusion until disease progression determined by investigator assessment of objective disease assessment per RECIST 1.1 .
Time to progression (TTP) outside the radiation field. | Assessed at week 6, 12, 24, 36, and 52.
  Defined as the time from inclusion until progression outside the radiation field determined by a CT, MR, or PET-CT per RECIST 1.1. Outside the radiation field is defined as outside and not adjacent to the PTV.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Felter, MD, Principal Investigator — Helev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Overeem Felter M, Moller PK, Josipovic M, Bekke SN, Bernchou U, Serup-Hansen E, Parikh P, Kim J, Geertsen P, Behrens CP, Madsen K, Vogelius IR, Topsoe JF, Berthelsen AK, Pohl M, Schytte T, Persson GF. 1-year efficacy results after MR-guided risk-adapted stereotactic radiotherapy of infra-diaphragmatic oligometastases in a multicenter phase II trial. Radiother Oncol. 2025 Apr;205:110748. doi: 10.1016/j.radonc.2025.110748. Epub 2025 Jan 27. PMID 39880308
- [Derived] van Overeem Felter M, Moller PK, Josipovic M, Bekke SN, Bernchou U, Serup-Hansen E, Madsen K, Parikh PJ, Kim J, Geertsen P, Behrens CP, Vogelius IR, Pohl M, Schytte T, Persson GF. MR-guided stereotactic radiotherapy of infra-diaphragmatic oligometastases: Evaluation of toxicity and dosimetric parameters. Radiother Oncol. 2024 Mar;192:110090. doi: 10.1016/j.radonc.2024.110090. Epub 2024 Jan 13. PMID 38224916